CLINICAL TRIAL: NCT01410734
Title: A Prospective Investigation of the Use of the Fluorescence Imaging on the da Vinci Surgical System for Intra-operative Near Infrared Imaging of the Biliary Tree
Brief Title: Fluorescence Imaging on the da Vinci Surgical System for Intra-operative Near Infrared Imaging of the Biliary Tree (up to 2-weeks Post-operatively)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intuitive Surgical (Industry)
Collaborators: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other); University Hospital, Geneva (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Fluorescence Bliliary ID
Record Dates: First submitted 2011-08-03; First posted 2011-08-05 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Gallbladder Disease; Biliary Colic; Gallstones
Keywords: cholecystectomy; chronic right upper quadrant pain
MeSH Terms: conditions — Gallbladder Diseases; Gallstones | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ICG (Experimental): Patient will received IV injection of ICG intra-operatively. Surgeon will view bile ducts under fluorescence imaging mode to see if ICG helps to identify biliary ducts.
  Interventions: Drug: Indocyanine green (ICG)

INTERVENTIONS:
Drug: Indocyanine green (ICG) — 2.5mg indocyanine green (ICG) will be administerly (IV injection) 30 minutes before surgery

SUMMARY:
The investigators hypothesize that the da Vinci Fluorescence Imaging Vision System provides real-time endoscopic near infrared fluorescence imaging of the biliary anatomy as defined as identifying biliary vessels; either cystic duct, common hepatic duct (CHD) or common bile duct (CBD). Irradiation given to the patient during a classic cholangiography can be reduced.

DETAILED DESCRIPTION:
Up to 40 patients will be prospectively enrolled in this multi-centre (up to 5 centres) single arm study. After given consent, patients will undergo minimally invasive cholecystectomy with da Vinci Fluorescence Imaging using Indocynine green (ICG) and near infra-red light (NIR) to identify the surgically relevant anatomy of the biliary tree during this procedure.

Efficacy endpoints The efficacy of the da Vinci Fluorescence Imaging Vision System to identify biliary anatomy will be demonstrated by successful detection (90%) of one or more of the following biliary vessels: Cystic duct, common hepatic duct (CHD) or common bile duct (CBD).

Safety endpoints To observe and report peri-operative safety outcomes, including but not limited to incidence of adverse events and allergic reactions (rare according to the current knowledge and applications). Safety endpoints will be met by affirming the safety profile of the procedure, compared to currently available literature.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Ages of 18 to 80 years.
* Symptoms consistent with gallbladder disease including biliary colic or chronic right upper quadrant pain.
* Ultrasound confirming gallstones

Exclusion Criteria:

* Acute cholecystitis
* Biliary pancreatitis
* Suspicion of common bile duct stones.
* Pregnancy.
* Previous upper abdominal open surgeries.
* Severe lack of cooperation by patient due to psychological or severe systemic illness.
* The presence of medical conditions contraindicating general anesthesia or standard surgical approaches.
* Subject has a previous history of adverse reaction or allergy to ICG, iodine products (or excipient), shellfish or iodine dyes
* Surgery converted to non-robotic procedures, such as open surgery or laparoscopic surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To identify biliary anatomy will be demonstrated by successful detection (90%) of one or more of the following biliary vessels: Cystic duct, common hepatic duct (CHD) or common bile duct (CBD). | intra-operatively

SECONDARY OUTCOMES:
observe and report peri-operative safety outcomes, including but not limited to incidence of adverse events and allergic reactions (rare according to the current knowledge and applications) | within 2 weeks post-operatively

CONTACTS AND LOCATIONS:
Locations (2):
- SS Antonio e Biagio e Cesare Arrigo, Alessandria, AL, Italy
- Hospital University Geneva, Geneva, Switzerland